CLINICAL TRIAL: NCT04725435
Title: Evaluation of Cerebral Oxygenation Results in Premature Infants: Kangaroo Care and Facilitated Tucking Example
Brief Title: Evaluation of Cerebral Oxygenation Results in Premature Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/42
Record Dates: First submitted 2021-01-15; First posted 2021-01-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Oxygenation; Premature; Kangaroo Care; Facilitated Tucking
Keywords: cerebral oxygenation; premature; kangaroo care; facilitated tucking
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: First sub purpose was designed as a single blind, parallel group, randomized controlled pre-test post-test order.
  Second sub purpose was designed as a single blind, parallel group, two intervention groups in pre-test and post-test order, and a randomized controlled control group.
Who Masked: Participant
Masking Description: Single (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo care (Experimental): No Intervention: Standard care The control group will be followed by infants using nesting in the incubator. It will be followed for 60 minutes without any action or application.
  Experimental: Kangaroo care The mother kangaroo will care for at least 60 minutes.
  Interventions: Behavioral: Kangaroo care
- Facilitated tucking position (Experimental): No Intervention: Standard care In the Control Group, the heel stick procedure will be performed in the infants own bed as in the clinical routine.
  Experimental 1: Manual Facilitated Tucking Position, infants will be given a manual facilitated tucking position during the heel stick procedure.
  Experimental 2: Facilitated Tucking Position, with the Nesting Bed (Tortoise Neo Bed), the facilitated tucking position will be given by the clinic nurse with the nesting bed during the heel stick collection procedure.
  Interventions: Behavioral: Facilitated Tucking Position

INTERVENTIONS:
Behavioral: Kangaroo care — Experimental: Kangaroo care The mother kangaroo will care for at least 60 minutes.
  Arms: Kangaroo care
Behavioral: Facilitated Tucking Position — Experimental 1: Manual Facilitated Tucking Position, infants will be given a manual facilitated tucking position during the heel stick procedure.
  Experimental 2: Facilitated Tucking Position with the Nesting Bed (Tortoise Neo Bed), the facilitated tucking position will be given by the clinic nurse with the nesting bed during the heel stick collection procedure.
  Arms: Facilitated tucking position

SUMMARY:
The general purpose of this project is; Evaluation of cerebral oxygenation results in premature infants.

These results will be evaluated in two different applications. The first practice and the first sub-aim of the study is to determine the effect of kangaroo care on cerebral oxygenation (rSO2) in premature infants.

The second application and purpose is to determine the effect of giving the infant the facilitated tucking position by hand and the nesting bed on the cerebral oxygenation (rSO2) of the infant during the heel blood collection process.

The study will be conducted between December 2020 and December 2021 at Level III NICU at the Medical Faculty Hospital in Konya.

DETAILED DESCRIPTION:
The general purpose of this project is; To determine the effect of kangaroo care and facilitated tucking position on cerebral oxygenation (rSO2) in premature infants.

In this context, the study has two sub-objectives. First sub purpose; to determine the effect of kangaroo care application given to premature inafants hospitalized in the NICU with the mother on cerebral oxygenation (rSO2), physiological parameters (heart rate, peripheral oxygen saturation (SpO2) and respiratory rate) and comfort / comfort levels.

This study was designed as a single blind, parallel group, pre-test and post-test randomized controlled trial.

First sub purpose; total sample size was determined as 40 preterm babies (20 in each group). Block randomization was used in this study. During the data collection phase, the purpose of the study will be explained to the parents of preterm infants by the researcher, and written consent will be obtained from the parents who agree to participate in the study through the "Informed Consent Form". Introductory Information Form, Physiological Parameter and rSO2 Follow-up Chart and Neonatal Comfort Scale created by the researcher will be used.

Second sub purpose; to determine the effect of facilitated tucking position on the infant's cerebral oxygenation (rSO2), physiological parameters (heart peak beat, SpO2 and respiratory rate), pain and comfort / comfort levels during the heel stick procedure.

This study was designed as a single blind, parallel group, two intervention groups in pre-test and post-test order, and a randomized controlled control group.

Second sub purpose; the total sample size was determined as 66 (22 in each group). Block randomization was used in this study. During the data collection phase, the purpose of the study will be explained to the parents of preterm infants by the researcher, and written consent will be obtained from the parents who agree to participate in the study through the "Informed Consent Form". The Introductory Information Form, Physiological Parameters and rSO2 Tracking Chart, PIPP-R and Neonatal Comfort Scale created by the researcher will be used.

ELIGIBILITY:
Inclusion Criteria:

* Adjusted gestational age of 28-36(+6) weeks at time of registration

Exclusion Criteria:

* Mechanical ventilation,
* Major congenital abnormalities,
* Surgical or severe medical morbidity (bronchopulmonary dysplasia, NEC, sepsis, or intraventricular bleeding)
* The mother is under 18 years of age
* The mother is not willing to do kangaroo care

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The first sub-purpose Outcome: rSO2 level | Change from baseline and 70 min
  Defines the change of rSO2 level. The NIRS monitor (COVIDEN Operations Manual INVOS® System, Model 5100C) was used to monitor rSO2 levels. The normal range of the rSO2 measured by the device was between 55% and 85%.
The first sub-purpose Outcome: physiological parameters of the premature infant- heart rate (min). | Change from baseline and 70 min
  Defines the change of heart rate (min) level.Philips IntelliVue MP40 device was used to monitor respiratory rate. Philips IntelliVue MP40 device was used to monitor heart rate (min).
The first sub-purpose Outcome: physiological parameters of the premature infant- SpO2 level | Change from baseline and 70 min
  Defines the change of SpO2 level.
The first sub-purpose Outcome: Neonates COMFORTneo scale | Change from baseline and 70 min
  The COMFORTneo scale is a Likert-type scale consisting of seven parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tonus. The items are rated between 0 and 10, and the score that can be obtained from the scale ranges between 6 and 30. A score of 4-6 indicates moderate pain and distress and that of 7-10 indicates severe pain and distress.
The first sub-purpose Outcome: physiological parameters of the premature infant-respiratory rate (min) | Change from baseline and 70 min
  Defines the change of respiratory rate (min) level.

SECONDARY OUTCOMES:
The second sub-purpose Outcome: Premature Infant Pain Profile Scale-Revised (PIPP-R) | Change from baseline and 70 min
  The PIPP-R scale includes 3 behavioral (frowning, squeezing eyes, nasolobial-groove), 2 physiological (heart rate and oxygen saturation) and 2 contextual (behavioral state and gestational age) items used in the assessment of pain in newborns. The items of the scale are scored as 3, 2, 1, 0 ((0-6 points that the pain is mild, 7-12 points is moderate, and 13-21 points is at a severe level.)
The second sub-purpose Outcome:Neonates The COMFORTneo Scale | Change from baseline and 70 min
  The scale consists of 7 items: muscle tone, alertness, facial tension, calmness / agitation, body movements, respiratory response, and crying. The lowest possible score from Newborn Comfort Behavior Scale is 6 and the highest score is 30. High scores indicate that the baby is not comfortable.
The second sub-purpose Outcome: physiological parameters of the premature infant- respiratory rate | Change from baseline and 70 min
  Defines the change of respiratory rate (min) level.
The second sub-purpose Outcome: physiological parameters of the premature infant- heart rate (min) | Change from baseline and 70 min
  Defines the change of heart rate (min) level.Philips IntelliVue MP40 device was used to monitor respiratory rate. Philips IntelliVue MP40 device was used to monitor heart rate (min).
The second sub-purpose Outcome: physiological parameters of the premature infant- oxygen saturation (%SpO2) | Change from baseline and 70 min
  Defines the change of SpO2 level.
The second sub-purpose Outcome: rSO2 level | Change from baseline and 70 min
  Defines the change of rSO2 level. The NIRS monitor (COVIDEN Operations Manual INVOS® System, Model 5100C) was used to monitor rSO2 levels. The normal range of the rSO2 measured by the device was between 55% and 85%.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Tas Arslan, Prof, Study Director — Selcuk University; Sibel Kucukoglu, assoc. prof., Study Director — Selcuk University; Deniz Kocoglu-Tanyer, assoc. prof., Study Chair — Selcuk University; Hanifi Soylu, Prof, Study Chair — Selcuk University; Murat Konak, assoc. prof., Study Director — Selcuk University; Sevinc Akkoyun, Msc, Study Director — Konya Ereğli State Hospital
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

REFERENCES:
- [Derived] Tas Arslan F, Akkoyun S, Kucukoglu S, Kocoglu-Tanyer D, Konak M, Soylu H. Effect of kangaroo mother care on cerebral oxygenation, physiological parameters, and comfort levels in late-premature infants: A randomized controlled trial. Midwifery. 2024 Oct;137:104096. doi: 10.1016/j.midw.2024.104096. Epub 2024 Jul 7. PMID 39024964